CLINICAL TRIAL: NCT00324922
Title: A Prospective, Randomized Trial Comparing Vancomycin With Trimethoprim/Sulfamethoxazole for the Treatment of MRSA Osteomyelitis
Brief Title: Vancomycin Or Trimethoprim/Sulfamethoxazole for Methicillin-resistant Staphylococcus Aureus Osteomyelitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Robert Harrington, Professor, Allergy & Infectious Diseases, Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27915
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Osteomyelitis; Methicillin-resistant Staphylococcus Aureus
Keywords: Vancomycin; Trimethoprim-Sulfamethoxazole Combination
MeSH Terms: conditions — Osteomyelitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Trimethoprim-sulfamethoxazole (Active Comparator): trimethoprim-sulfamethoxazole, double strength, 2-3 tabs twice a day by mouth for 6-12 weeks
  Interventions: Drug: trimethoprim-sulfamethoxazole; Drug: vancomycin
- Vancomycin (Active Comparator): Vancomycin, dosage to be determined by serum levels, medication provided by vein and duration 6-12 weeks
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole — trimethoprim/sulfamethoxazole 320/1600 mg po bid
  Arms: Trimethoprim-sulfamethoxazole
Drug: vancomycin — 1g iv bid

SUMMARY:
The primary question of this study is to understand if trimethoprim-sulfamethoxazole (TMP-SMX) is as effective as vancomycin for treating methicillin-resistant Staphylococcus aureus (MRSA) osteomyelitis.

DETAILED DESCRIPTION:
Treatment of osteomyelitis is hampered by a paucity of evidence from prospective clinical trials with randomized treatment arms. Furthermore, previous randomized or observational trials have enrolled small numbers of subjects and thus often had non-definitive findings. One of the most common causes of osteomyelitis is Staphylococcus aureus. Over the past 10 years, rates of methicillin-resistant S. aureus (MRSA) have risen dramatically. Vancomycin is currently the treatment of choice for treating MRSA. While vancomycin is effective, it is only available in intravenous formulation and has renal and bone marrow toxicities. There is a critical need for effective, oral, cheap drugs for the treatment of MRSA. Trimethoprim-sulfamethoxazole (TMP-SMX) is a drug with several advantageous properties for the treatment of MRSA osteomyelitis. To address this question regarding optimal treatment of MRSA osteomyelitis, we designed a prospective, randomized trial comparing TMP-SMX with vancomycin for the treatment of MRSA osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

1. Culture-proven MRSA, obtained in operating room or sterile biopsy procedure from bone site. The infection and sampling site can either be within bone or a deep soft-tissue site that is contiguous with bone; OR radiographic abnormality consistent with osteomyelitis in conjunction with a positive blood culture for MRSA.
2. Surgical debridement of infection site, as needed.
3. Subject is capable of providing written informed consent.
4. Subject is at least 18 years of age.
5. Subject capable of receiving outpatient parenteral therapy for 12 weeks.

Exclusion Criteria:

1. Hypersensitivity to TMP-SMX or vancomycin.
2. S. aureus resistant to TMP-SMX or vancomycin.
3. Osteomyelitis that develops directly from a chronic, open wound.
4. Polymicrobial culture(the only exception is if coagulase-negative staphylococcus is present in the culture and the clinical assessment is that it is a contaminant).
5. Subject has a positive pregnancy test at study enrollment.
6. Convicted felon currently in prison.
7. Baseline renal or hepatic insufficiency that would preclude administration of study drugs.
8. Active injection drug use without safe conditions to administer intravenous antibiotics for 3 months.
9. Anticipated use of antibiotics for greater than 14 days for an infection other than osteomyelitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2006-05-01 (Actual); Primary Completion 2007-05-01 (Actual); Study Completion 2007-05-01 (Actual)

PRIMARY OUTCOMES:
Clinical cure | 12 months
  No clinical or radiographic evidence of infection at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy H. Dellitt, MD, Principal Investigator — UW; Jeanne Chan, PharmD, MPH, Principal Investigator — UW; Matthew Golden, MD, MPH, Principal Investigator — UW; M. Bradford Henley, MD, Principal Investigator — UW; Jeanne M Marrazzo, MD, MPH, Principal Investigator — UW; Lisa Taitsman, MD, Principal Investigator — UW; Thomas R Hawn, MD, PhD, Principal Investigator — UW; Robert D Harrington, MD, Principal Investigator — UW; Christian Ramers, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States